CLINICAL TRIAL: NCT02903147
Title: The Efficacy of a Functional Meta-Cognitive Intervention to Improve Human Factors of Professional Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Navah Ratzon, Professor, Occupational Therapist, Tel Aviv University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rachel Shichrur; Navah Ratzon (Other: Pricipal Investigator, Prof)
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Human Risk Factors; Driving Behavior; Meta-cognition
Keywords: IVDR; driving behavior patterns; Meta-Cognitive Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Meta-Cognitive Intervention (Experimental): The intervention is aimed to improve human factors of professional bus drivers
  Interventions: Behavioral: Functional Meta-Cognitive Intervention
- Control group (Active Comparator): The control group had the employer's training - The company holds routine covert inspections, summons to conversations with the security offices and records in the drivers' personal files.
  Interventions: Behavioral: The employer's training

INTERVENTIONS:
Behavioral: Functional Meta-Cognitive Intervention — Functional-Meta-Cognitive Intervention Program was focused on raising awareness to safe driving risk factors identified at pre-screening, with reference to the difficulties that the driver raises and providing coping strategies. The intervention has been customized for each driver and included three sessions of two hours.
  Arms: Functional Meta-Cognitive Intervention
Behavioral: The employer's training
  Arms: Control group

SUMMARY:
The objective of the study is to examine the effectiveness of a functional-meta-cognitive intervention program to reduce driving risk factors amongst professional bus drivers.

DETAILED DESCRIPTION:
In Israel, the percentage of professional drivers involved in lethal car accidents is high in relation to their number on the roads. Every car accident involving a bus driver could potentially put at risk the lives of tens of passengers, and cause damages both direct and indirect at high costs. Due to the high risk of the bus drivers and their passengers, it is highly important to identify and improve the driving characteristics which are necessary for safer driving of said drivers. Many studies have assessed and identified the risk factors of safe driving, but there is relatively little research-based evidence concerning the ability to improve the driving skills of drivers in general and in particular of bus drivers, which are considered a high risk group.

According to the National Road Safety Authority, 88% of road accidents are caused by driver errors. Therefore, the real challenge is to provide a better understanding in the role of human factors in causing road accidents to try and develop a variety of effective interventions to reduce these risk factors. This understanding can contribute both to a better assessment of professional drivers' driving fitness and to intervene accordingly. In this study, we have focused on main aspects that exist in relevant literature and are human risk factors: Cognitive-perceptual, ergonomic and personality risk factors, and checked the connection between these risk factors and actual monitored driving scores as recorder by an In-Vehicle Data Recorder (IVDR). In addition, we examined the effectiveness of a functional-meta-cognitive intervention program designed to increase drivers' awareness to their way of driving. The research model is based on previous driving models and the guiding occupational therapy practice framework model in Israel, while adjusting the model to the professional driving in public transportation line of work and its particular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Male gender.
* Having a valid bus driver's license.
* Working for a specific large bus company in the center of Israel.

Exclusion Criteria:

* Drivers who had less than 50 hours of IVDR data were excluded.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in In Vehicle Data Recorder (IVDR) risk score | Change from baseline IVDR risk score at 1 year
  Assessing the degree of change in the rate of IVDR events before and after intervention.

SECONDARY OUTCOMES:
Change in car accident rate | Change from ratings of questionnaire pre intervention to ratings at an average of 1 year post intervention.
  Assessing the change in the rate of accidents per year before and after the intervention in the intervention group.
Change in subjective ratings of driving performance questionnaire. | Change from ratings of questionnaire at baseline pre intervention to reratings at an average of 1 year post intervention..
  Assessing the change in the subjective ratings of the level of performance and of satisfaction with performance before and after the intervention in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Navah Ratzon, Prof., Principal Investigator — Tel Aviv University

IPD SHARING:
Plan to Share IPD: Undecided